CLINICAL TRIAL: NCT00794287
Title: Performance of CAST (Cellular Antigen Stiumulation Test)in Patients With Wasp Venom Allergy. Evaluation of Neutralizing IgG Subclasses
Brief Title: Performance of CAST (Cellular Antigen Stimulation Test) in Patients With Wasp Venom Allergy: Evaluation of Neutralizing IgG Subclasses
Status: Withdrawn | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: PD Dr. Thomas Kündig, University of Zurich
Other Study IDs: ZU-AgNT-004
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Wasp Venom Allergic Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Hymenoptera allergic patients before allergen specific immunotherapy
  Interventions: Other: Taking blood samples
- 2: Hymenoptera allergic patients after allergen specific immunotherapy
  Interventions: Other: Taking blood samples

INTERVENTIONS:
Other: Taking blood samples — No intervention is done. Only blood samples are taken.

SUMMARY:
To determine which subclass of IgG in the serum of patients undergoing SIT against wasp venom is able to neutralize the allergen, and therefore to prevent a positive CAST

ELIGIBILITY:
Inclusion criteria:

* male and female patient with allergy to wasp venom grade III and IV according to H.L. Müller
* 18-75 years
* planned SIT against wasp venom or finished 5 years SIT against wsp venom (10/10)

Exclusion criteria:

* oral corticosteroids
* chromogycin
* ketotifen
* immunosuppressive drugs within the last 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wasp venom allergic patients grade III and IV according to H.L. Müller in the age group of 18-75 years
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland